CLINICAL TRIAL: NCT02351609
Title: Patient Navigation and Financial Incentives to Promote Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Karen Lasser, BMC Faculty, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-3296; 125785-RSG-14-034-01CPPB (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; patient navigation; financial incentives; health disparities
MeSH Terms: conditions — Smoking Cessation | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients in this arm will receive a low literacy smoking cessation educational brochure and a list of resources for smoking cessation. Patients will also receive navigation from a trained navigator Patients will receive up to 4 hours of patient navigation, in person or over the phone, over a 6-month period. Patients will receive financial incentives for biochemically confirmed smoking cessation.
  Interventions: Behavioral: Intervention
- Enhanced Traditional Care control (Active Comparator): Patients receive information about smoking cessation resources and an educational brochure developed by the Massachusetts Department of Public Health.
  Interventions: Other: Enhanced Traditional Care control

INTERVENTIONS:
Behavioral: Intervention — Intervention patients will be introduced to the patient navigator either in person or by telephone. The intervention patients will receive navigation from one of two trained navigators, based centrally in the Section of General Internal Medicine. The purpose of the patient navigation interactions is to 1) connect patients to existing yet underutilized smoking cessation resources and 2) increase patient commitment to follow through with existing treatment services.
  Financial incentives: $250 for biochemically confirmed abstinence within six months after study enrollment, and $500 for biochemically confirmed abstinence for an additional six months after the initial cessation.
  Arms: Intervention
Other: Enhanced Traditional Care control — List of smoking cessation resources and educational brochure.
  Arms: Enhanced Traditional Care control

SUMMARY:
Cigarette smoking is a significant health threat. To eliminate disparities in cancer burden, smoking rates must be reduced among populations where smoking is disproportionately concentrated: those with low socioeconomic status (SES). The investigators will apply two methods that are being used in the field of health disparities to the challenge of promoting smoking cessation among low SES smokers. These include: 1) Patient navigation; patient navigators are often lay persons, working as paid employees, who guide patients through the health care system and 2) Financial incentives; investigators propose to provide monetary incentives: $250 for smoking cessation within 6 months after study enrollment, and $500 for an additional 6 months of abstinence after the initial cessation. The investigators will recruit/randomize 352 smokers to a randomized controlled trial comparing the combination of Patient Navigation (delivered over 6 months) and Financial Incentives versus Enhanced Traditional Care control condition (smoking cessation brochure/list of cessation resources). The RCT will take place among adult daily smokers seen in the past year at BMC primary care practices, with a primary outcome of smoking cessation at one year. Follow-up by telephone, for both groups, will occur 6, 12, and 18 months after enrollment.

DETAILED DESCRIPTION:
Cigarette smoking is a highly significant health threat, responsible for > 480,000 deaths in the US each year, many due to cancer, and is the largest cause of preventable morbidity and mortality in the US. Primary care settings provide an opportunity to reach large proportions of low-income smokers, as 61% of such smokers are engaged in medical care. The proposed project addresses this under-utilization of available smoking cessation services which is occurring despite considerable interest among low-income patients about quitting/receiving help with quitting. This intervention has the potential to increase the reach of existing services and in turn, to improve the public's health.

Patient financial incentives, while not yet used as standard of care for health promotion, are in the research stage for various types of conditions. Financial incentives are effective in promoting smoking cessation; but have not been extensively studied among low SES smokers. Financial incentives are a behavioral economic intervention that is effective in promoting smoking cessation, increasing cessation rates 3-fold compared to no incentives. The investigators believe financial incentives merit further study, particularly in low SES populations. Incentives for completing smoking cessation programs/achieving abstinence may be particularly effective among low SES smokers because they: 1) can alleviate some of the financial strain that prevents low SES smokers from quitting (studies have shown that the stress from financial problems prevents patients from quitting, even though quitting smoking could save people large amounts of money); 2) promote short-term abstinence among smokers with mental illness and substance use, many of whom are low SES smokers; 3) provide a substitute reinforcer for smoking (e.g., in lieu of hobbies, physical activity, work satisfaction) often absent in environments of low SES smokers and 4) provide extrinsic motivation for patients to quit smoking, and may be particularly effective among low SES smokers, many of whom in our recent pilot study were found to have low levels of intrinsic motivation. Our strategy is to combine financial incentives with patient navigation, as the latter may "supercharge" the former, for the two interventions may work in complementary ways. The investigators posit that incentives will augment people's willingness to connect with a navigator, and the navigator will put people in touch with resources/environments in which the incentives can work.

Patient navigation holds promise as an intervention to reduce cancer disparities, but alone may be insufficient to promote smoking cessation. Patient navigators are often lay persons from the community who guide patients through the health care system so that they receive appropriate services. While patient navigation has been shown to be an effective intervention to reduce health care disparities, prior patient navigation studies have been limited to the realms of cancer screening and diagnosis. Preliminary findings from our pilot RCT of patient navigation to promote smoking cessation among low SES and minority primary care patients at Boston Medical Center suggest that a more potent intervention may be needed. While a patient navigator was able to link 37% of patients to treatment, she was unable to contact or meaningfully connect with 53% of patients. Thus, financial incentives may be used to increase participant motivation to connect with patient navigators.

Combining financial incentives with patient navigation may be an effective approach to promote cessation among low SES and minority smokers. Multicomponent interventions have shown the most promise in changing health behaviors in general, and in reducing health disparities. Barriers to behavior change among socially disadvantaged persons may be so large that no single intervention can be effective. The investigators have therefore chosen to implement two intervention components, financial incentives and patient navigation, which have shown some promise in smoking cessation, and are currently being applied in the health disparities field to other health conditions.

Our objectives and hypotheses are:

Specific Aim I: To determine whether patient navigation and financial incentives increase the rates at which primary care patients engage in smoking cessation treatment.

H1: Compared to control patients, those assigned to the intervention will be more likely to engage in smoking cessation treatment at six months post-enrollment.

Specific Aim II: To determine whether patient navigation and financial incentives increase the rates at which primary care patients quit smoking (our primary outcome), defined as biochemically confirmed cessation at twelve months using salivary cotinine levels.

H1: Compared to ETC patients, those assigned to the patient navigation/financial incentives intervention will be more likely to be abstinent at 12 months post-enrollment.

ELIGIBILITY:
Inclusion Criteria:

(1) age ≥ 18; (2) smoked ≥10 cigarettes/day in the past week; (3) have a scheduled visit with a PCP at BMC on the day of enrollment or within the next six months; (4) telephone access (5) English speaking; (6) plan on quitting smoking within the next six months; (7) able and willing to participate in the study protocol and provide informed consent.

Exclusion Criteria:

(1) planning to move out of the area within the next six months; (2) cognitive impairments that preclude participation in study activities; (3) severe illness or distress; (4) inability to read/understand English; (5) actively using evidence-based smoking cessation treatment; (6) transient residence or lack of a telephone for follow-up assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-03-03 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence at 12 months post-enrollment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen Lasser, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Abidoye O, Ferguson MK, Salgia R. Lung carcinoma in African Americans. Nat Clin Pract Oncol. 2007 Feb;4(2):118-29. doi: 10.1038/ncponc0718. PMID 17259932
- [Background] Yancy CW. Executive summary of the African-American Initiative. MedGenMed. 2007 Feb 8;9(1):28. PMID 17435635
- [Background] Kurian AK, Cardarelli KM. Racial and ethnic differences in cardiovascular disease risk factors: a systematic review. Ethn Dis. 2007 Winter;17(1):143-52. PMID 17274224
- [Background] Unger B, Kemp JS, Wilkins D, Psara R, Ledbetter T, Graham M, Case M, Thach BT. Racial disparity and modifiable risk factors among infants dying suddenly and unexpectedly. Pediatrics. 2003 Feb;111(2):E127-31. doi: 10.1542/peds.111.2.e127. PMID 12563085
- [Background] Cokkinides VE, Halpern MT, Barbeau EM, Ward E, Thun MJ. Racial and ethnic disparities in smoking-cessation interventions: analysis of the 2005 National Health Interview Survey. Am J Prev Med. 2008 May;34(5):404-12. doi: 10.1016/j.amepre.2008.02.003. PMID 18407007
- [Background] Volpp KG, Troxel AB, Pauly MV, Glick HA, Puig A, Asch DA, Galvin R, Zhu J, Wan F, DeGuzman J, Corbett E, Weiner J, Audrain-McGovern J. A randomized, controlled trial of financial incentives for smoking cessation. N Engl J Med. 2009 Feb 12;360(7):699-709. doi: 10.1056/NEJMsa0806819. PMID 19213683
- [Background] Higgins ST, Alessi SM, Dantona RL. Voucher-based incentives. A substance abuse treatment innovation. Addict Behav. 2002 Nov-Dec;27(6):887-910. doi: 10.1016/s0306-4603(02)00297-6. PMID 12369474
- [Background] Van Etten ML, Higgins ST, Budney AJ, Badger GJ. Comparison of the frequency and enjoyability of pleasant events in cocaine abusers vs. non-abusers using a standardized behavioral inventory. Addiction. 1998 Nov;93(11):1669-80. doi: 10.1046/j.1360-0443.1998.931116695.x. PMID 9926530
- [Background] Higgins ST, Bickel WK, Hughes JR. Influence of an alternative reinforcer on human cocaine self-administration. Life Sci. 1994;55(3):179-87. doi: 10.1016/0024-3205(94)00878-7. PMID 8007760
- [Background] Audrain-McGovern J, Rodriguez D, Epstein LH, Rodgers K, Cuevas J, Wileyto EP. Young adult smoking: what factors differentiate ex-smokers, smoking cessation treatment seekers and nontreatment seekers? Addict Behav. 2009 Dec;34(12):1036-41. doi: 10.1016/j.addbeh.2009.06.012. Epub 2009 Jul 5. PMID 19619948
- [Background] Chin MH, Walters AE, Cook SC, Huang ES. Interventions to reduce racial and ethnic disparities in health care. Med Care Res Rev. 2007 Oct;64(5 Suppl):7S-28S. doi: 10.1177/1077558707305413. PMID 17881624
- [Background] Donatelle RJ, Prows SL, Champeau D, Hudson D. Randomised controlled trial using social support and financial incentives for high risk pregnant smokers: significant other supporter (SOS) program. Tob Control. 2000;9 Suppl 3(Suppl 3):III67-9. doi: 10.1136/tc.9.suppl_3.iii67. No abstract available. PMID 10982912
- [Background] Shoptaw S, Jarvik ME, Ling W, Rawson RA. Contingency management for tobacco smoking in methadone-maintained opiate addicts. Addict Behav. 1996 May-Jun;21(3):409-12. doi: 10.1016/0306-4603(95)00066-6. PMID 8883490
- [Background] Dohan D, Schrag D. Using navigators to improve care of underserved patients: current practices and approaches. Cancer. 2005 Aug 15;104(4):848-55. doi: 10.1002/cncr.21214. PMID 16010658
- [Background] Lasser KE, Murillo J, Medlin E, Lisboa S, Valley-Shah L, Fletcher RH, Emmons KM, Ayanian JZ. A multilevel intervention to promote colorectal cancer screening among community health center patients: results of a pilot study. BMC Fam Pract. 2009 May 29;10:37. doi: 10.1186/1471-2296-10-37. PMID 19480698
- [Background] Percac-Lima S, Grant RW, Green AR, Ashburner JM, Gamba G, Oo S, Richter JM, Atlas SJ. A culturally tailored navigator program for colorectal cancer screening in a community health center: a randomized, controlled trial. J Gen Intern Med. 2009 Feb;24(2):211-7. doi: 10.1007/s11606-008-0864-x. PMID 19067085
- [Background] Fang CY, Ma GX, Tan Y, Chi N. A multifaceted intervention to increase cervical cancer screening among underserved Korean women. Cancer Epidemiol Biomarkers Prev. 2007 Jun;16(6):1298-302. doi: 10.1158/1055-9965.EPI-07-0091. PMID 17548702
- [Background] Battaglia TA, Roloff K, Posner MA, Freund KM. Improving follow-up to abnormal breast cancer screening in an urban population. A patient navigation intervention. Cancer. 2007 Jan 15;109(2 Suppl):359-67. doi: 10.1002/cncr.22354. PMID 17123275
- [Background] Wang C, Burris MA. Photovoice: concept, methodology, and use for participatory needs assessment. Health Educ Behav. 1997 Jun;24(3):369-87. doi: 10.1177/109019819702400309. PMID 9158980
- [Background] Hergenrather KC, Rhodes SD, Cowan CA, Bardhoshi G, Pula S. Photovoice as community-based participatory research: a qualitative review. Am J Health Behav. 2009 Nov-Dec;33(6):686-98. doi: 10.5993/ajhb.33.6.6. PMID 19320617
- [Background] Catalani C, Minkler M. Photovoice: a review of the literature in health and public health. Health Educ Behav. 2010 Jun;37(3):424-51. doi: 10.1177/1090198109342084. Epub 2009 Oct 1. PMID 19797541
- [Background] DiMatteo MR, Giordani PJ, Lepper HS, Croghan TW. Patient adherence and medical treatment outcomes: a meta-analysis. Med Care. 2002 Sep;40(9):794-811. doi: 10.1097/00005650-200209000-00009. PMID 12218770
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Kanner AD, Coyne JC, Schaefer C, Lazarus RS. Comparison of two modes of stress measurement: daily hassles and uplifts versus major life events. J Behav Med. 1981 Mar;4(1):1-39. doi: 10.1007/BF00844845. PMID 7288876
- [Background] Romano PS, Bloom J, Syme SL. Smoking, social support, and hassles in an urban African-American community. Am J Public Health. 1991 Nov;81(11):1415-22. doi: 10.2105/ajph.81.11.1415. PMID 1951797
- [Background] Klesges RC, Brown K, Pascale RW, Murphy M, Williams E, Cigrang JA. Factors associated with participation, attrition, and outcome in a smoking cessation program at the workplace. Health Psychol. 1988;7(6):575-89. doi: 10.1037//0278-6133.7.6.575. PMID 3215163
- [Background] Curry SJ, Marlatt GA, Gordon J, Baer JS. A comparison of alternative theoretical approaches to smoking cessation and relapse. Health Psychol. 1988;7(6):545-56. doi: 10.1037//0278-6133.7.6.545. PMID 3215161
- [Background] Centers for Disease Control and Prevention (CDC). State-specific secondhand smoke exposure and current cigarette smoking among adults - United States, 2008. MMWR Morb Mortal Wkly Rep. 2009 Nov 13;58(44):1232-5. PMID 19910910
- [Background] Volpp KG, John LK, Troxel AB, Norton L, Fassbender J, Loewenstein G. Financial incentive-based approaches for weight loss: a randomized trial. JAMA. 2008 Dec 10;300(22):2631-7. doi: 10.1001/jama.2008.804. PMID 19066383
- [Background] Sorensen G, Barbeau E, Hunt MK, Emmons K. Reducing social disparities in tobacco use: a social-contextual model for reducing tobacco use among blue-collar workers. Am J Public Health. 2004 Feb;94(2):230-9. doi: 10.2105/ajph.94.2.230. PMID 14759932
- [Background] Lasser K, Boyd JW, Woolhandler S, Himmelstein DU, McCormick D, Bor DH. Smoking and mental illness: A population-based prevalence study. JAMA. 2000 Nov 22-29;284(20):2606-10. doi: 10.1001/jama.284.20.2606. PMID 11086367
- [Background] Emmons KM, Stoddard AM, Fletcher R, Gutheil C, Suarez EG, Lobb R, Weeks J, Bigby JA. Cancer prevention among working class, multiethnic adults: results of the healthy directions-health centers study. Am J Public Health. 2005 Jul;95(7):1200-5. doi: 10.2105/AJPH.2004.038695. Epub 2005 Jun 2. PMID 15933240
- [Background] Lai DT, Cahill K, Qin Y, Tang JL. Motivational interviewing for smoking cessation. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD006936. doi: 10.1002/14651858.CD006936.pub2. PMID 20091612
- [Background] Gilpin EA, Pierce JP, Farkas AJ. Duration of smoking abstinence and success in quitting. J Natl Cancer Inst. 1997 Apr 16;89(8):572-6. doi: 10.1093/jnci/89.8.572. PMID 9106646
- [Background] Abrams DB, Follick MJ, Biener L, Carey KB, Hitti J. Saliva cotinine as a measure of smoking status in field settings. Am J Public Health. 1987 Jul;77(7):846-8. doi: 10.2105/ajph.77.7.846. PMID 3592039
- [Background] Caraballo RS, Giovino GA, Pechacek TF, Mowery PD, Richter PA, Strauss WJ, Sharp DJ, Eriksen MP, Pirkle JL, Maurer KR. Racial and ethnic differences in serum cotinine levels of cigarette smokers: Third National Health and Nutrition Examination Survey, 1988-1991. JAMA. 1998 Jul 8;280(2):135-9. doi: 10.1001/jama.280.2.135. PMID 9669785
- [Background] Jarvis MJ, Tunstall-Pedoe H, Feyerabend C, Vesey C, Saloojee Y. Comparison of tests used to distinguish smokers from nonsmokers. Am J Public Health. 1987 Nov;77(11):1435-8. doi: 10.2105/ajph.77.11.1435. PMID 3661797
- [Background] Condiotte MM, Lichtenstein E. Self-efficacy and relapse in smoking cessation programs. J Consult Clin Psychol. 1981 Oct;49(5):648-58. doi: 10.1037//0022-006x.49.5.648. No abstract available. PMID 7287974
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Zhu SH, Anderson CM, Tedeschi GJ, Rosbrook B, Johnson CE, Byrd M, Gutierrez-Terrell E. Evidence of real-world effectiveness of a telephone quitline for smokers. N Engl J Med. 2002 Oct 3;347(14):1087-93. doi: 10.1056/NEJMsa020660. PMID 12362011
- [Background] An LC, Zhu SH, Nelson DB, Arikian NJ, Nugent S, Partin MR, Joseph AM. Benefits of telephone care over primary care for smoking cessation: a randomized trial. Arch Intern Med. 2006 Mar 13;166(5):536-42. doi: 10.1001/archinte.166.5.536. PMID 16534040
- [Background] Crawford SL, Tennstedt SL, McKinlay JB. A comparison of anlaytic methods for non-random missingness of outcome data. J Clin Epidemiol. 1995 Feb;48(2):209-19. doi: 10.1016/0895-4356(94)00124-9. PMID 7869067
- [Background] Deci EL, Koestner R, Ryan RM. A meta-analytic review of experiments examining the effects of extrinsic rewards on intrinsic motivation. Psychol Bull. 1999 Nov;125(6):627-68; discussion 692-700. doi: 10.1037/0033-2909.125.6.627. PMID 10589297
- [Background] Centers for Disease Control and Prevention (CDC). State-specific smoking-attributable mortality and years of potential life lost--United States, 2000-2004. MMWR Morb Mortal Wkly Rep. 2009 Jan 23;58(2):29-33. PMID 19165137
- [Background] Kanjilal S, Gregg EW, Cheng YJ, Zhang P, Nelson DE, Mensah G, Beckles GL. Socioeconomic status and trends in disparities in 4 major risk factors for cardiovascular disease among US adults, 1971-2002. Arch Intern Med. 2006 Nov 27;166(21):2348-55. doi: 10.1001/archinte.166.21.2348. PMID 17130388
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Lasser KE, Quintiliani LM, Truong V, Xuan Z, Murillo J, Jean C, Pbert L. Effect of Patient Navigation and Financial Incentives on Smoking Cessation Among Primary Care Patients at an Urban Safety-Net Hospital: A Randomized Clinical Trial. JAMA Intern Med. 2017 Dec 1;177(12):1798-1807. doi: 10.1001/jamainternmed.2017.4372. PMID 29084312